CLINICAL TRIAL: NCT05089981
Title: The Efficacy and Safety of N-acetyl-L-cysteine (NAC) as Adjuvant Therapy in Acute on Chronic Liver Failure (ACLF) A Randomized Double Blind Placebo Controlled Pilot Trial
Brief Title: Intravenous NAC Use in ACLF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: National Institute of Liver & GI Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Syed Hasnain Ali Shah, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-1245-13480
Record Dates: First submitted 2021-09-29; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Acute on Chronic Liver Failure(ACLF)
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC group (Active Comparator): IV N acetyl cysteine 300mg will be administered in doses as described in protocol
  Interventions: Drug: N acetyl cysteine
- NAC Placebo group (Placebo Comparator): IV Placebo of N acetyl cysteine will be administered in doses as described in protocol (Placebo will be normal saline in a look alike preparation with same volume as active NAC arm)
  Interventions: Drug: Placebo of N acetyl cysteine

INTERVENTIONS:
Drug: N acetyl cysteine — Intravenous use of N acetyl cysteine in prescribed doses
  Arms: NAC group
Drug: Placebo of N acetyl cysteine — Intravenous Placebo of N Acetyl cysteine in look alike form (Normal saline)
  Arms: NAC Placebo group

SUMMARY:
Primary Objective To evaluate the efficacy and safety of 72 hour NAC treatment regimen in the management of ACLF

Secondary Objective To evaluate the six weeks mortality and length of hospital stay in ACLF patients treated with NAC

Randomized, Double blind pilot study of IV N-Acetyl cysteine for the treatment of ACLF. Participants will be randomized into intervention and control arm using block randomization by computer generated random numbers. Efficacy will be assessed by clinical improvement in symptoms and signs of decompensated chronic liver disease (CLD). To assess safety degree of adverse reactions will be observed. Periodic assessments until 28 day will be done consisting of Physical exam, safety assessments, vital signs and lab tests.

Dose of Drug: 72 hour regimen consisting of three doses of intravenous N-Acetyl cysteine will be used for a total dose of 300mg/kg.

Number of Patients: 100 Accrual period: 15 months

DETAILED DESCRIPTION:
Introduction:

Acute on Chronic Liver Failure (ACLF) is a relatively new entity, characterized by complications of cirrhosis and high rate of organ failures. Short term mortality at 28 days is high (>15%). ACLF is multifactorial in its etiology and there is no consensus about the definitions between different parts of the world. The Asian Pacific Association for the Study of the Liver (APASL) consensus defines ACLF as "Acute hepatic insult manifesting as jaundice (serum bilirubin ≥ 5mg/dl and coagulopathy (INR≥1.5 or prothrombin activity <40% complicated within 4 weeks by clinical ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease or cirrhosis, and is associated with a high 28-day day mortality. Another definition of ACLF defines it as "an acute deterioration of pre-existing chronic liver disease, usually related to a precipitating event and associated with increased mortality at 3 months due to multi-system organ failure". This definition also includes a high mortality at 28 days and organ failures.

Events known to precipitate ACLF include Acute alcoholic hepatitis, acute hepatotrophic viral infections , reactivation of hepatitis B virus infection, Drug induced liver injury (DILI), Gastrointestinal bleeding, sepsis, ischemia to the liver and portal vein thrombosis.

An enhanced pro-inflammatory cytokine environment has been shown to be present in ACLF. These are chronically primed neutrophils which are energy depleted and unable to carry out the phagocytosis function, leading to a functional failure in combating infections.

Cytokines also play a key role in the pathogenesis of the inflammatory response. Elevated serum levels of TNF-α, sTNF-αR1, sTNF-αR2, interleukin (IL)-2, IL-2R, IL-4, IL-6, IL-6,IL-8, IL-10 and interferon-γ have been described. Raised levels of these pro-inflammatory cytokines can be due to necrotic liver cells, reduced clearance by the liver or most importantly, from activation of toll-like receptors (TLRs). These receptors activate Kupffer cells (KCs), which play a key role I the pathogenesis of liver injury by activating signaling cascades, transcription of pro-inflammatory cytokines and super oxide agents. The resulting oxidative stress releases proteolytic enzymes and vasoactive substances like endothelin-1 (ET-1), thromboxane A2, nitric oxide (NO), and prostaglandins which lead to microcirculatory dysfunction. The entire cascade ultimately results in hepatocyte death and liver dysfunction.

The reactive oxygen species (ROS) released by kupffer cells activate hepatic stellate cells (HSCs) leading to increased synthesis of extracellular matrix (ECM). Oxidative stress (OS) leads to worsening inflammation, focal and zonal necrosis in the liver and thus architectural distortion. Several studies relating to liver diseases indicate an over production of ROS and/or reduction of hepatic Gutathione (GSH) which is the most abundant cellular anti-oxidant, which exhibits numerous and versatile functions and therefore protects cells against toxicity regardless of etiology of disease. N-Acetyle cystein (NAC) has an optimal thiol redox state, which helps protective ability of the cell to counter balance OS and inflammation. NAC has been used in a variety of clinical conditions, such as inflammatory bowel disease, pulmonary diseases, cystic fibrosis, septic shock and aceto-aminophen and non-aceto-aminophen induced acute liver failure (ALF). Moreover, it has also been found to improve liver blood flow and liver function in septic shock and non-alcoholic fatty liver disease.

Methodology:

Trial design The study is a randomized double blind placebo controlled pilot trial. Study Settings The trial will be conducted in in-patient units of Aga Khan University Hospital (AKUH) & National Institute of Liver Diseases (NILGID), Dow university Hospital where ACLF patients are admitted. Patients will be followed up for survival six weeks post discharge.

Study population:

Inclusion criteria:

* Patients with ACLF having CLIF-C ACLF (Acute-on-Chronic Liver Failure) scores of 35 to 65 will be enrolled in this study.
* Establishment of ACLF grade 1-3 according to EASL- CLIFF criteria
* Willing to provide informed consent to participate in the study (by study subject or next of kin)

Exclusion criteria:

* History of hypersensitivity to NAC
* Hepatocellular carcinoma
* Pregnancy
* Advanced cardiovascular, neurological or pulmonary disease

Subject Screening and Recruitment:

The patients admitted with ACLF at the two sites will be enrolled in this study. Clinical and laboratory criteria will establish the diagnosis of ACLF.

Randomization and Allocation:

Two treatments of A, B and Block size of 2 x 2= 4 Concealed allocation is assured by using of a central web-based system. A double-dummy design would be implemented for subject and study personnel blinding. Blinded assessors will collect outcomes data.

Blinding:

The study will be double blinded to avoid any biases. Participant as well as investigators will be blinded to the intervention assignment. The assignment will be kept in concealed envelopes.

Group I:

Intravenous N-acetylcysteine in standard IV form. Infusion of NAC shall be administered as follows:

72 hour regimen: consists of 3 doses; total dose delivered: 300 mg/kg Loading dose: 150 mg/kg (maximum 15 g) infused over 60 minutes Second dose: 50 mg/kg (max 5g) infused over 4 hours Third dose: 100mg/kg (maximum: 10 g) infused over 67 hours Patients will be monitored for 96 hours post treatment.

Group II:

Patient in this arm will be treated with standard of care and will receive identical placebo in IV form for 72 hours additionally.

Composition: Normal saline with identical color and package

Methods and assessments

Laboratory assessments required:

* Complete blood count
* Prothrombin time ratio, APTT, INR
* Blood urea nitrogen
* Serum creatinine levels
* Liver function profile including total protein group
* Oxygen saturation
* Abdominal ultrasound
* Albumin
* Procalcitonin
* CRP
* Arterial ammonia
* Interleukin-10
* TNF- alpha
* ABGs
* Lactate
* Blood random glucose
* Oxidized albumin

Subject Compliance Monitoring:

Random checks will be done by the PI and team to ensure protocol compliance.

Study Duration:

The total duration of study is 15 months. Each participant will be follow up to 6 weeks (+/- 7 days). The study will be closed when required number of participants and follow-up time has been completed or participants have documented events.

Discontinuation criteria:

* Liver transplant
* Death
* sever adverse reaction

An interim-analysis will be perform on the primary endpoint when 25% of patients have been randomized and have completed the 6 weeks follow-up

Any SAE which develop within 24 hours of completion of NAC infusion will be considered as treatment emergent.

Safety reporting:

Investigators and study team will be monitor and reporting the adverse event/reaction during the study trial through online pharmacy ADR form

serious adverse events (SAE):

Respectively, any adverse event or adverse reaction that:

* results in death
* is life-threatening*
* requires hospitalisation or prolongation of existing hospitalisation**
* results in persistent or significant disability or incapacity
* consists of a congenital anomaly or birth defect
* other important medical event(s)***

Referrences:

1. Moreau R, Arroyo Vincente. Acute-on-Chronic Liver Failure: A new clinical entity. Clinical Gastroenterology and Hepatology 2015;13: 836-841
2. Sarin S et al. Acute-on chronic liver failure:consensus recommendations of the Asia Pacific association for the study of the liver (APASL). Hepatol Int. 2014;8:453-471
3. Moreau R et al. Acute-on chronic liver failure is a distinct syndrome which develops in patients with acute decompensation of cirrhosis. Gastroenterology 2013;144: 1426-1437
4. Arroyo V, Moreau R, Lalan R. et al. Acute-0on-chronic liver failure: A new syndrome that will re-classify cirrhosis. J Hepatology 2015;62: S131-S143
5. Sarin S, Choudhary A, Acute-on-chronic liver failure: terminology, mechanisms and management: Nature reviews: Gastroenterology and Hepatology 2016
6. Asrani SK, O'Leary JG, Acute-on-chronic liver failure. Clin Liver Dis 2014;18: 561-574
7. Jalan R, Gines P, Olson JC et al. Acute-on-chronic liver failure. J Hepatol 2012;57:1336-1348
8. Gustot T. Multiple organ failure in sepsis: prognosis and role of systemic inflammatory response. Curr opin Crit care.2011;17:153-159
9. Sen S, Davies NA, Mookerjee RP et al. Pathophysiological effect of albumin dialysis in acute-on-chronic liver failure: a randomized controlled study. Liver Transpl 2004;10: 1109-1119
10. Bilzer M, Roggel F,Gerbes AL, Role of Kupffer cells in host defense and liver disease. Liver Int 2006; 26: 1175-1186 Holland-Fischer P, Gronbaek H, Sandhl TD et al. Kupffer cells are activated in cirrhotic portal hypertension and not normalized by TIPS. Gut 2011;60: 1389-139315 months
11. The Efficacy and safety of N-acetyl-L-cysteine (NAC) as adjuvant therapy in acute on chronic liver failure (ACLF)
12. A randomized double blind placebo controlled pilot trial

14. Rockey DC, Fouasier L, Chung JJ, et al. Cellular localization of of endothelin-1 and increased production of liver injury in the rat potential for autocrine and paracrine effects on stellate cells. Hepatology 1998;27: 472-480 15. Diesen DL, Kuo PC, Nitric Oxide and redox regulaton in the liver Part 11. Redox biology in pathologic hepatocytes and implications for intervention. J Surg Res 2011; 167, 96-112 16. Chatterjee R, Mitra A, An overview of effective therapies and recent advances in biomarkers for chronic liver disease and associated cancer. Int. Immunopharmacol 2015; 24: 335-345 17. Mussaco-Sebio R, Saporito-Magrina C,Semprine J et al, J Inorg Biochem 2014; 137: 94-100 18. Okanoue T, Mitsuyoushi H. Non-alcoholic steatohepatitis,oxdative stress and NASH. Nihon Naika Gakkai Zasshi 2006, 95,51-56 19. Kersksick C, Willoughby D, The anti-oxidant role of Glutathione and N-acetylcysteine supplements and exercise induced oxidative stress. J Int Soc Sports Nutrition 2005;9: 38-44 20. Moura FA, de Andrale KQ, Dos Santos JC, et al. Anti-oxidant therapy for the treatment of inBa-Ma pigflammatory bowel disease: Does it work? Redox Biol 2015; 6: 617-639 21. Li J, Zhang S, Wu Y, Protective effects of N-acetylcysteine on the liver of brain dead mini pig. Transplant Proc 2010: 42: 195-199

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion will be

  * Age between 18 and 70 years
  * Establishment of ACLF grade 1-3 according to EASL- CLIFF criteria
  * Willing to provide informed consent to participate in the study (by study subject or next of kin)

Exclusion Criteria:

* Criteria for exclusion will be

  * History of hypersensitivity to NAC
  * Hepatocellular carcinoma
  * pregnancy
  * Advanced cardiovascular or pulmonary disease
  * Advanced primary neurological disease (such as stroke)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy & safety of NAC in the improvement of ACLF To evaluate the efficacy and safety of 72 hour NAC treatment regimen in the management of ACLF | 72 hrs
  clinical and biochemical improvement will be noted as NAC efficacy and safety through AE & SAE

SECONDARY OUTCOMES:
6-weeks Survival | 6 weeks
  A 6-weeks survival data will be collected for this secondary outcome measure
Length of hospital stay | 6 weeks
  Length of hospital stay in patients treated with NAC Vs Placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University,, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No